CLINICAL TRIAL: NCT00442741
Title: An Open Label Phase I Study to Evaluate the Effects of Patupilone on the Pharmacokinetics of Midazolam and Omeprazole in Patients With Advanced Malignancies (Extension)
Brief Title: Evaluate the Effects of Patupilone on the Pharmacokinetics of Midazolam and Omeprazole in Patients With Advanced Malignancies (Extension)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: pts. will be captured in core
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2123E1
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Solid Tumors
Keywords: Cancer; EPO906; Patupilone
MeSH Terms: conditions — Neoplasms | interventions — epothilone B; Omeprazole

ARMS (2):
- Patupilone + Midazolam (Experimental)
  Interventions: Drug: Patupilone
- Patupilone + Omeprazole (Experimental)
  Interventions: Drug: Patupilone + Omeprazole

INTERVENTIONS:
Drug: Patupilone
  Arms: Patupilone + Midazolam
Drug: Patupilone + Omeprazole
  Arms: Patupilone + Omeprazole

SUMMARY:
The purpose of this extension study is to evaluate the potential inhibitory effects of patupilone on metabolism using midazolam and omeprazole as the respective probe drugs.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients 18 years or older
* Histologically documented advanced solid tumor, who have failed standard systemic therapy, or for whom standard systemic therapy does not exist
* Completed the Core study
* Completed all sampling in the core and not dose reduced Patients with adequate hematologic parameters

Exclusion criteria:

* Female patients who are pregnant or breast-feeding.
* Patients with a severe and/or uncontrolled medical disease
* Patients with a known diagnosis of human immunodeficiency virus (HIV) infection
* Patients having received an investigational agent within 30 days prior to study entry

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and potential activity of patupilone once every 21 days in patients that completed the core study

SECONDARY OUTCOMES:
Assessment of objective response and tumor evaluation will be based on the response evaluation criteria in solid tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals